CLINICAL TRIAL: NCT00132366
Title: Cortical Excitability in Succinic Semialdehyde Dehydrogenase Deficiency
Brief Title: Brain Excitability in Patients With Succinic Semialdehyde Dehydrogenase Deficiency
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050224; 05-N-0224
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-06-25

CONDITIONS: Succinic Semialdehyde; Dehydrogenase Deficiency; Diseases
Keywords: Neurotransmission; Cortical Excitability; GABA; Seizures; Succinic Semialdehyde Dehydrogenase Deficiency; SSADH; Healthy Volunteer; HV
MeSH Terms: conditions — Disease; Seizures; succinic semialdehyde dehydrogenase deficiency

SUMMARY:
This study will measure brain excitability in patients with succinic semialdehyde dehydrogenase (SSADH) deficiency, and in their parents. SSADH is a rare inherited disease in which changes in certain brain chemicals affect brain cell activity. Symptoms vary greatly among patients, and may include mental retardation, impaired ability to coordinate movements, and delays in language and speech development. Other symptoms may include poor muscle tone, uncontrolled seizures and other neurological or behavioral abnormalities. Test findings in patients and their parents will be compared with those of healthy normal volunteers.

The following individuals may be eligible for this study: patients with SSADH who are between 5 and 24 years of age; parents of patients who are between 18 and 55 years of age; healthy normal children who are between 10 and 17 years of age; and healthy normal adults who are between 18 and 55 years of age. Candidates are screened with blood and urine tests.

All participants undergo the following:

* Transcranial magnetic stimulation (TMS): This procedure maps brain function. A wire coil is held on the scalp, and a brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions to help position the coil properly. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the subject may hear a click and feel a pulling sensation on the skin under the coil. During the test, electrical activity of muscles is recorded with a computer or other recording device, using electrodes attached to the skin with tape.
* Magnetic resonance imaging (MRI): This test combines a powerful magnet with an advanced computer system and radio waves to produce accurate, detailed pictures of organs and tissues. During the scan, the subject lies on a table in a narrow cylinder containing a magnetic field, wearing ear plugs to muffle loud noises that occur with electrical switching of the magnetic fields. He or she can speak with a staff member via an intercom system at all times during the procedure. In addition to standard MRI, subjects may have newer MRI tests, such as diffusion tensor MRI and magnetic resonance spectroscopy.

In addition to the above, patients and their parents may also undergo the following tests:

* Electroencephalography (EEG): This test records brain waves (electrical activity of the brain). Electrodes are placed on the scalp and brain electrical activity is recorded while the subject lies quietly, breathes deeply, watches flashes of light, or sleeps. Some patients may also have video-EEG monitoring, which involves simultaneous clinical recording using a video camera along with brain wave recording.
* Sleep study and multiple sleep latency onset testing (MSLT): Electrodes are placed on the subject's scalp and remain there while the subject sleeps in the hospital overnight. MSLT is done the next day, starting 2 hours after the subject wakes up from the night's sleep. A total of five 20- to 30-minute naps are recorded, each every 2 hours, to access daytime sleepiness.
* Nerve conduction studies: This test measures the speed with which nerves conduct electrical impulses and the strength of the connection between the nerve and the muscle. A probe is placed on the skin to deliver a small electrical stimulus, and wires taped on the skin record the impulses.

DETAILED DESCRIPTION:
Objective: To study cortical excitability, electroencephalography patterns, nerve conduction velocity, and sleep patterns, in succinic semialdehyde dehydrogenase (SSADH) deficiency, a rare autosomal recessive pediatric neurotransmitter disease associated with elevated levels of brain gamma aminobutyric acid (GABA), the major inhibitory neurotransmitter. The clinical phenotype includes mental retardation, epilepsy, and neuropsychiatric manifestations.

Study Population: Patients with SSADH deficiency, parents of patients (who are obligate heterozygotes), and healthy volunteers.

Design: This is a natural history study in which subjects will have a series of neurophysiological tests. Transcranial magnetic stimulation (TMS) is a non-invasive technique that allows for measures of cortical excitation and inhibition. Electroencephalography (EEG) measures baseline brain electrical activity. Nerve conduction studies measure the speed of conduction of impulses by peripheral nerves. Polysomnography records sleep cycles and associated eye movements, muscle potentials, heart rate, and respiration.

Outcome measures: Motor cortex excitability threshold, paired pulse facilitation, and paired pulse inhibition on TMS will be the main outcome measures. Values will be compared across the 4 groups of patients, carriers, adult and child healthy volunteers. Additional measures will include nerve conduction velocity, EEG frequency, and sleep patterns.

ELIGIBILITY:
* INCLUSION CRITERIA

Patients

* Persistent 4-hydroxybutyric aciduria (gamma-hydroxybutyric aciduria)
* Documented succinic semialdehyde dehydrogenase enzyme deficiency
* English-speaking (or the ability to understand English as a second language)
* Patients must have clinically documented SSADH deficiency.
* Patients may be male or female.
* Female patients of child bearing potential will have a pregnancy test prior to the study to ensure that pregnant patients will not participate in the study.
* During the study, women of child bearing potential must use a reliable method of birth control.

Patients will be aged 5-24

Parents will be aged 18-55

Adult Healthy Volunteers will be aged 18-55

Child Healthy Volunteers will be aged 10-17

EXCLUSION CRITERIA

* Major debilitating mental or physical illness that would interfere with participation.
* Pregnancy or lactation
* Use of alcohol or recreational drugs during the study
* Patients with progressive neurologic disorders
* Patients with a history of significant medical disorders
* Patients requiring treatment of drugs known to affect the GABAergic system, including vigabatrin.
* Patients with cancer.
* Patients who had seizure activity 24 hours prior to the study.

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2005-08-16; Primary Completion 2008-06-30 (Actual); Study Completion 2008-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Akaboshi S, Hogema BM, Novelletto A, Malaspina P, Salomons GS, Maropoulos GD, Jakobs C, Grompe M, Gibson KM. Mutational spectrum of the succinate semialdehyde dehydrogenase (ALDH5A1) gene and functional analysis of 27 novel disease-causing mutations in patients with SSADH deficiency. Hum Mutat. 2003 Dec;22(6):442-50. doi: 10.1002/humu.10288. PMID 14635103
- [Background] Arnold S, Berthele A, Drzezga A, Tolle TR, Weis S, Werhahn KJ, Henkel A, Yousry TA, Winkler PA, Bartenstein P, Noachtar S. Reduction of benzodiazepine receptor binding is related to the seizure onset zone in extratemporal focal cortical dysplasia. Epilepsia. 2000 Jul;41(7):818-24. doi: 10.1111/j.1528-1157.2000.tb00248.x. PMID 10897152
- [Background] Bonham JR, Downing M, Pollitt RJ, Manning NJ, Carpenter KH, Olpin SE, Allen JC, Worthy E. Quality assessment of urinary organic acid analysis. Ann Clin Biochem. 1994 Mar;31 ( Pt 2):129-33. doi: 10.1177/000456329403100203. PMID 8060090